CLINICAL TRIAL: NCT04362072
Title: Single-Arm Study of Lorlatinib in Participants With Anaplastic Lymphoma Kinase (ALK)-Positive Non-Small Cell Lung Cancer (NSCLC) Whose Disease Progressed After One Prior Second-Generation ALK Tyrosine Kinase Inhibitor (TKI)
Brief Title: Study of Lorlatinib In People With ALK-positive Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7461027; 2019-002504-41 (EudraCT Number)
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Carcinoma; Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma | interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lorlatinib (Experimental): Participants will take 100 mg (four, 25 mg tablets) once daily.
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — 25 milligram (mg) tablet

SUMMARY:
The purpose of this clinical trial is to learn whether the study medicine (called lorlatinib) is safe and effective for the treatment of non-small cell lung cancer that is caused by an abnormal anaplastic lymphoma kinase (ALK) gene.

This study is seeking participants whose lung cancer has progressed after receiving either alectinib or ceritinib as their first treatment.

Participants will take part in this study for up to approximately 4 years, depending on when the study is completed and how their cancer responds to the study treatment. They will take lorlatinib orally (by mouth) once daily.

Participants will visit the study site about every six weeks to meet with the study team. During these visits, the study team will monitor the safety and effects of lorlatinib.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have evidence of histologically or cytologically confirmed diagnosis of metastatic NSCLC (Stage IV, American Joint Committee on Cancer [AJCC] v7.0) that carries an ALK rearrangement.
* Disease Status Requirements: disease progression after alectinib or ceritinib as first line therapy (the study will limit enrollment of participants with best response of progression or indeterminate on prior alectinib to 8 participants). Participants may have had prior chemotherapy, but only if before starting treatment with alectinib or ceritinib.
* Tumor Requirements: All Participants must have at least one measurable target extracranial lesion according to RECIST v1.1. Participants with asymptomatic CNS metastases (including participants controlled with stable or decreasing steroid use within the last 2 weeks prior to study entry) will be eligible. Participants who have leptomeningeal disease (LM) or carcinomatous meningitis (CM) will be eligible if the LM/CM is visualized on magnetic resonance imaging (MRI) or if documented baseline cerebral spinal fluid (CSF) positive cytology is available.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
* Adequate bone marrow functioning, pancreatic function, renal function and liver function
* Acute effects of any prior therapy resolved to baseline severity or to CTCAE Grade ≤1 except for adverse events (AEs) that in the investigator' judgment do not constitute a safety risk for the participant.
* Systemic anti-cancer therapy with alectinib or ceritinib discontinued within a minimum of 5 half-lives prior to first dose of lorlatinib on the study (unless clinically meaningful tumor flare per discretion of the investigator, in which discussion with the sponsor is warranted).
* Male participants are eligible to participate if they agree to use proper contraception during the intervention period and for at least 98 days after the last dose of study intervention
* Female participants are eligible to participate if they are not pregnant or breastfeeding, and agree to use proper contraception during the intervention period and for at least 35 days after the last dose of study intervention.
* Capable of giving signed informed consent and willingness and ability to comply with the study scheduled visits and other procedures.

Exclusion criteria:

* Prior ALK TKI treatment or anti-cancer treatment other than first line alectinib or ceritinib.
* Spinal cord compression unless the participant has good pain control attained through therapy, and there is stabilization or recovery of neurological function for the 4 weeks prior to randomization.
* Gastrointestinal abnormalities, including inability to take oral medication; requirement for intravenous alimentation; prior surgical procedures affecting absorption including total gastric resection or lap band; active inflammatory gastrointestinal disease, chronic diarrhea, symptomatic diverticular disease; treatment for active peptic ulcer disease in the past 6 months; malabsorption syndromes.
* Active and clinically significant bacterial, fungal, or viral infection including hepatitis B virus (HBV) or hepatitis C virus (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS) related illness.
* Clinically significant vascular (both arterial and venous) and non-vascular cardiac conditions, (active or within 3 months prior to enrollment)
* Participants presenting with abnormal Left Ventricular Ejection Fraction (LVEF) by echocardiogram or Multi-Gated Acquisition Scan according to institutional lower limits.
* Participants with predisposing characteristics for acute pancreatitis according to investigator judgment
* History or known presence of interstitial fibrosis, interstitial lung disease, pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis, and pulmonary fibrosis.
* Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Evidence of active malignancy (other than current NSCLC, non-melanoma skin cancer, in situ cervical cancer, papillary thyroid cancer, ductal carcinoma in situ (DCIS) of the breast or localized and presumed cured prostate cancer) within the last 3 years prior to randomization.
* Radiation therapy (except palliative to relieve bone pain) within 2 weeks of study entry. Palliative radiation must have been completed at least 48 hours prior to study entry. Stereotactic or small field brain irradiation must have completed at least 2 weeks prior to study entry. Whole brain radiation must have completed at least 4 weeks prior to study entry.
* Prior irradiation to >25% of the bone marrow.
* Concurrent use of any of the following food or drugs within 12 days prior to the first dose of lorlatinib: known strong CYP3A inducers, known strong CYP3A inhibitors, known CYP3A substrates with narrow therapeutic index, known permeability glycoprotein (P-gp) substrates with a narrow therapeutic index
* Major surgery within 4 weeks prior to enrollment.
* Known prior or suspected severe hypersensitivity to study interventions or any component in their formulations.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- UCI Medical Center/Chao Family Comprehensive Cancer Center, Orange, California, United States
- India (4):
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, DEL
  - Healthcare Global Enterprises, Bengaluru, Karnataka
  - Bhakti Vedanta Hospital and Research Institute, Thane, Maharashtra
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
- Italy (8):
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, MI
  - Centro Riferimento Oncologico di Aviano - IRCCS SOC Oncologia Medica e dei Tumori Immunocorrelati, Aviano, PN
  - Azienda Ospedaliero Universitaria di Parma, Parma, PR
  - Azienda Ospedaliera San Camillo Forlanini, Roma, ROME
  - AOU San Luigi Gonzaga, Orbassano (TO), TO
  - AO Santa Maria della Misericordia, Perugia, Umbria
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
- Poland (5):
  - Ms Pneumed Janusz Milanowski, Katarzyna Szmygin-Milanowska Spolka Jawna, Lublin
  - Centrum Medyczne EVOMED, Szczecin
  - Dom Lekarski Centrum Medyczne Outlet Park, Szczecin
  - Pracownia Medycyny Nuklearnej, 109 Szpital Wojskowy z Przychodnia SP ZOZ, Szczecin
  - Dom Lekarski S.A., Szczecin
- Spain (8):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Teresa Herrera (C.H.U.A.C), A Coruña
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - ICO L'Hospitalet (Hospital Duran i Reynals), L'Hospitalet de Llobregat
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Kantonsspital Graubuenden, Chur, Kanton Graubünden, Switzerland
- United Kingdom (3):
  - Guy's and St Thomas' NHS Foundation Trust, London
  - NIHR/Wellcome Trust Clinical Research Facility, Manchester
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461027

RESULTS

PARTICIPANT FLOW:
Groups:
- Lorlatinib: Participants received Lorlatinib 100 milligrams (mg) (25 mg*4 tablets) orally once daily (QD) in 21-day cycles. Participants continued to receive study treatment until objective disease progression, unacceptable toxicity, participant refusal, lost to follow up or death, whichever occurred first.
Period: Treatment
Arm/Group | Lorlatinib
Started | 71
Completed | 0
Not Completed | 71
Not completed — Adverse Event | 1
Not completed — Death | 9
Not completed — Physician Decision | 2
Not completed — Progressive disease | 27
Not completed — Withdrawal by Subject | 4
Not completed — Global deterioration of health status | 1
Not completed — Switched to commercial Lorlatinib | 13
Not completed — Entered Lorlatinib continuation Study | 11
Not completed — Other | 3
Period: Follow up
Arm/Group | Lorlatinib
Started | 35
Completed | 31
Not Completed | 4
Not completed — Death | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Groups:
- Lorlatinib: Participants received Lorlatinib 100 mg (25 mg*4 tablets) orally QD in 21-day cycles. Participants continued to receive study treatment until objective disease progression, unacceptable toxicity, participant refusal, lost to follow up or death, whichever occurred first.
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.14 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 15
  Race: White | 54
  Race: Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed Overall Objective Response (OR) as Per Independent Central Review (ICR) as Assessed by RECIST v1.1
Description: Confirmed OR based on ICR assessment was defined as complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumor (RECIST) version(v)1.1 from date of first dose until documented progressive disease (PD) or start of new anti-cancer therapy without regard to discontinuation from treatment. Both CR and PR must be confirmed by repeat assessments performed no less than 4 weeks after criteria for response are first met. CR: disappearance of all target and non-target lesions. PR: at least 30 % decrease in sum of diameters of target, taking as reference baseline sum diameters. PD: at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 millimeter (mm). Appearance of one or more new lesions was also considered sign of progression. For non-target PD: unequivocal progression of existing non-target lesions.
Time Frame: From date of first dose until documented PD or start of new anti-cancer therapy, whichever occurred earlier (maximum treatment exposure up to 42.78 months)
Population: Intent to treat (ITT) analysis population included all enrolled participants who took at least 1 dose of Lorlatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Percentage of participants | 42.3 [30.6 to 54.6]

2. Secondary Outcome: Percentage of Participants With Confirmed OR as Per Investigator (INV) as Assessed by RECIST v 1.1
Description: Confirmed OR based on derived investigator assessment was defined as CR or PR according to RECIST v1.1 from date of first dose until PD or start of new anti-cancer therapy without regard to discontinuation from treatment. Both CR and PR must be confirmed by repeat assessments performed no less than 4 weeks after criteria for response are first met. CR: disappearance of all target and non-target lesions. PR: at least 30 % decrease in sum of diameters of target, taking as reference baseline sum diameters. PD: at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered sign of progression. For non-target PD: unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 1
Population: ITT analysis population included all enrolled participants who took at least 1 dose of Lorlatinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Percentage of participants | 36.6 [25.5 to 48.9]

3. Secondary Outcome: Percentage of Participants With Confirmed Intracranial (IC) Objective Response (IC-OR) as Per ICR as Assessed by RECIST v 1.1
Description: IC-OR based on ICR assessment was defined as IC-CR or PR according to RECIST v1.1 from date of first dose until documented IC-PD or start of new anti-cancer therapy without regard to discontinuation from treatment. Both IC-CR and IC-PR must be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response are first met. CR: disappearance of all target and non-target lesions. PR: at least 30 % decrease in sum of diameters of target, taking as reference baseline sum diameters. PD: at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered sign of progression. For non-target PD: unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 1
Population: Per-protocol analysis population based on ICR (PPICR) included all enrolled participants who took at least 1 dose of Lorlatinib and had central nervous system (CNS) metastases at study entry (i.e. with lesions having disease site = brain) according to ICR.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 30
Percentage of participants | 46.7 [28.3 to 65.7]

4. Secondary Outcome: Percentage of Participants With Confirmed IC-OR as Per INV as Assessed by RECIST v 1.1
Description: IC-OR based on derived investigator assessment was defined as IC-CR or PR according to RECIST v1.1 from date of first dose until documented IC-PD or start of new anti-cancer therapy without regard to discontinuation from treatment. Both IC-CR and IC-PR must be confirmed by repeat assessments performed no less than 4 weeks after the criteria for response are first met. CR: disappearance of all target and non-target lesions. PR: at least 30 % decrease in sum of diameters of target, taking as reference baseline sum diameters. PD: at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered sign of progression. For non-target PD: unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 1
Population: Per-protocol analysis population based on (PPINV) included all enrolled participants who took at least 1 dose of Lorlatinib and had CNS metastases at study entry (i.e. with lesions having disease site = brain) according to investigator.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 23
Percentage of participants | 56.5 [34.5 to 76.8]

5. Secondary Outcome: Time to Response (TTR) as Per ICR as Assessed by RECIST v 1.1
Description: TTR based on ICR assessments was defined, for participants with a confirmed OR, as the time from the date of first dose to the first documentation of OR (CR or PR) which was subsequently confirmed. For participants whose OR proceeded from PR to CR, the onset of PR was taken as the onset of response. CR: disappearance of all target and non-target lesions. PR: at least 30 % decrease in sum of diameters of target, taking as reference baseline sum diameters.
Time Frame: From date of first dose until first documented objective response, CR or PR (maximum treatment exposure up to 42.78 months)
Population: Analysis population included all enrolled participants who took at least 1 dose of Lorlatinib and had confirmed CR or PR as per ICR.
Measure: Median (Full Range); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 30
Months | 1.5 [1.2 to 8.4]

6. Secondary Outcome: TTR as Per INV as Assessed by RECIST v 1.1
Description: TTR based on derived investigator assessments was defined, for participants with a confirmed objective response, as the time from the date of first dose to the first documentation of objective response (CR or PR) which is subsequently confirmed. For participants whose OR proceeds from PR to CR, the onset of PR is taken as the onset of response. CR: disappearance of all target and non-target lesions. PR: at least 30 % decrease in sum of diameters of target, taking as reference baseline sum diameters.
Time Frame: as for outcome 5
Population: Analysis population included all enrolled participants who took at least 1 dose of Lorlatinib and had confirmed CR or PR as per INV.
Measure: Median (Full Range); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 26
Months | 1.6 [1.2 to 8.3]

7. Secondary Outcome: Duration of Response (DOR) as Per ICR as Assessed by RECIST v 1.1
Description: DOR: for participants with confirmed OR per ICR, as time from first documentation of OR (CR/PR whichever was earlier) to date of first documentation of PD/death due to any cause, whichever occurred first. CR:disappearance of all target and non-target lesions. PR:at least 30 % decrease in sum of diameters of target, taking as reference baseline sum diameters. PD:at least 20% increase in sum of diameters of target lesions,taking as reference smallest sum on study. Addition to relative increase of 20%, sum must also demonstrate absolute increase of at least 5mm. Appearance of one/ more new lesions: sign of progression. For non-target PD:unequivocal progression of existing non-target lesions. Participants who completed/discontinued study without PD/death, as well as who received alternate anti-cancer therapy prior to PD, were censored at their last adequate response assessment date/last adequate assessment prior to start date of alternate anti-cancer therapy. Analysis:Kaplan-Meier method.
Time Frame: From first documented OR (CR or PR) to date of first documented PD or death due to any cause or censoring date, whichever occurred first (maximum treatment exposure up to 42.78 months)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 30
Months | NA [8.6 to NA] — Median and upper limit of 95% confidence interval (CI) is not estimable due to insufficient data.

8. Secondary Outcome: DOR as Per INV as Assessed by RECIST v 1.1
Description: DOR: for participants with confirmed OR per investigator,as time from first documentation of OR(CR/PR whichever was earlier) to date of first documentation of PD/death due to any cause, whichever occurred first. CR:disappearance of all target and non-target lesions. PR:at least 30% decrease in sum of diameters of target,taking as reference baseline sum diameters. PD:at least 20% increase in sum of diameters of target lesions,taking as reference smallest sum on study. Addition to relative increase of 20%,sum must also demonstrate absolute increase of at least 5mm. Appearance of one/more new lesions:sign of progression. For non-target PD:unequivocal progression of existing non-target lesions. Participants who completed/discontinued study without PD/death,as well as who received alternate anti-cancer therapy prior to PD,were censored at their last adequate response assessment date/last adequate assessment prior to start date of alternate anti-cancer therapy. Analysis:Kaplan-Meier method.
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 26
Months | 20.9 [9.9 to NA] — Upper limit of 95% CI is not estimable due to insufficient data.

9. Secondary Outcome: Duration of Intracranial Response (IC-DoR) as Per ICR as Assessed by RECIST v 1.1
Description: IC-DoR: for participants with confirmed objective intra-cranial response per ICR, as time from first documentation of objective intra-cranial response (CR/PR whichever is earlier) to date of first documentation of PD in brain or death due to any cause, whichever occurs first. CR: disappearance of all target and non-target lesions. PR: at least 30 % decrease in sum of diameters of target, taking as reference baseline sum diameters. PD: at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. Appearance of one/more new lesions:sign of progression. For non-target PD: unequivocal progression of existing non-target lesions. Participants who completed or discontinued study without PD or death, as well as participants who received alternate anti-cancer therapy prior to PD, were censored at their last adequate response assessment date or last adequate assessment prior to start date of alternate anti-cancer therapy. Analysis: Kaplan-Meier method.
Time Frame: From first documented IC-OR (CR or PR) to date of first documented PD or death due to any cause or censoring date, whichever occurred first (maximum treatment exposure up to 42.78 months)
Population: Per-protocol analysis population based on ICR (PPICR) included all enrolled participants who took at least 1 dose of Lorlatinib and had central nervous system (CNS) metastases at study entry (i.e. with lesions having disease site = brain) according to ICR. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 14
Months | NA [NA to NA] — Median, upper and lower limit of 95% CI is not estimable due to insufficient data.

10. Secondary Outcome: IC-DoR as Per INV as Assessed by RECIST v 1.1
Description: IC-DoR: for participants with confirmed objective intra-cranial response, per investigator as time from first documentation of objective intra-cranial response (CR or PR whichever is earlier) to date of first documentation of PD in brain or death due to any cause, whichever occurs first. CR: disappearance of all target and non-target lesions. PR: at least 30 % decrease in sum of diameters of target, taking as reference baseline sum diameters. PD: at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. Appearance of one/more new lesions: sign of progression. For non-target PD: unequivocal progression of existing non-target lesions. Participants who completed or discontinued study without PD or death, as well as who received alternate anti-cancer therapy prior to PD, were censored at their last adequate response assessment date or last adequate assessment prior to start date of alternate anti-cancer therapy. Analysis: Kaplan-Meier method.
Time Frame: as for outcome 9
Population: Per-protocol analysis population based on (PPINV) included all enrolled participants who took at least 1 dose of Lorlatinib and had CNS metastases at study entry (i.e. with lesions having disease site = brain) according to investigator. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 13
Months | NA [NA to NA] — Median, upper and lower limit of 95% CI is not estimable due to insufficient data.

11. Secondary Outcome: Time to Tumor Progression (TTP) as Per ICR as Assessed by RECIST v 1.1
Description: TTP according to RECIST v1.1 as time from date of first dose to the date of the first documentation of PD per IRC. PD was defined as at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered sign of progression. For non-target PD: unequivocal progression of existing non-target lesions. Participants who completed or discontinued study without PD or death, as well as participants who received alternate anti-cancer therapy prior to PD, were censored at their last adequate response assessment date or last adequate assessment prior to start date of alternate anti-cancer therapy. Analysis was performed using Kaplan-Meier method.
Time Frame: From date of first dose until first documented PD or censoring date, whichever occurred first (maximum treatment exposure up to 42.78 months)
Population: ITT analysis population included all enrolled participants who took at least 1 dose of Lorlatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Months | 18.0 [9.7 to NA] — Upper limit of 95% CI is not estimable due to insufficient data.

12. Secondary Outcome: TTP as Per INV as Assessed by RECIST v 1.1
Description: TTP according to RECIST v1.1 as time from date of first dose to the date of the first documentation of PD per investigator. PD was defined as at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered sign of progression. For non-target PD: unequivocal progression of existing non-target lesions. Participants who completed or discontinued study without PD or death, as well as participants who received alternate anti-cancer therapy prior to PD, were censored at their last adequate response assessment date or last adequate assessment prior to start date of alternate anti-cancer therapy. Analysis was performed using Kaplan-Meier method.
Time Frame: as for outcome 11
Population: ITT analysis population included all enrolled participants who took at least 1 dose of Lorlatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Months | 12.2 [8.3 to 24.8]

13. Secondary Outcome: Progression-Free Survival (PFS) as Per ICR as Assessed by RECIST v 1.1
Description: PFS according to RECIST v1.1 was defined as the time from date of first dose to the date of the first documentation of PD per ICR or death due to any cause, whichever occurred first. PD was defined as at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered sign of progression. For non-target PD: unequivocal progression of existing non-target lesions. Participants who completed or discontinued study without PD or death, as well as participants who received alternate anti-cancer therapy prior to PD, were censored at their last adequate response assessment date or last adequate assessment prior to start date of alternate anti-cancer therapy. Analysis was performed using Kaplan-Meier method.
Time Frame: From date of first dose until first documented PD or death or censoring date, whichever occurred first (maximum treatment exposure up to 42.78 months)
Population: ITT analysis population included all enrolled participants who took at least 1 dose of Lorlatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Months | 12.2 [6.9 to 22.1]

14. Secondary Outcome: PFS as Per INV as Assessed by RECIST v 1.1
Description: PFS according to RECIST v1.1 was defined as the time from date of first dose to the date of the first documentation of PD per investigator or death due to any cause, whichever occurred first. PD was defined as at least 20% increase in sum of diameters of target lesions, taking as reference smallest sum on study. In addition to relative increase of 20%, sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions was also considered sign of progression. For non-target PD: unequivocal progression of existing non-target lesions. Participants who completed or discontinued study without PD or death, as well as participants who received alternate anti-cancer therapy prior to PD, were censored at their last adequate response assessment date or last adequate assessment prior to start date of alternate anti-cancer therapy. Analysis was performed using Kaplan-Meier method.
Time Frame: as for outcome 13
Population: ITT analysis population included all enrolled participants who took at least 1 dose of Lorlatinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Months | 9.7 [6.9 to 18.4]

15. Secondary Outcome: Time to Intra-Cranial Response (IC-TTR) as Per ICR as Assessed by RECIST v 1.1
Description: IC-TTR: for participants with a confirmed IC-OR per ICR, was defined as the time from the date of first dose to the first documentation of objective intra-cranial response (CR or PR) which is subsequently confirmed. For participants whose IC-OR proceeds from PR to CR, the onset of PR was taken as the onset of response. CR: disappearance of all target and non-target lesions. PR: at least 30 % decrease in sum of diameters of target, taking as reference baseline sum diameters.
Time Frame: From date of first dose to the first documented objective intra-cranial response (CR or PR) (maximum treatment exposure up to 42.78 months)
Population: PPICR included all enrolled participants who took at least 1 dose of Lorlatinib and had central nervous system (CNS) metastases at study entry (i.e. with lesions having disease site = brain) according to ICR. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 14
Months | 2.8 [1.3 to 12.6]

16. Secondary Outcome: IC-TTR as Per INV as Assessed by RECIST v 1.1
Description: IC-TTR: for participants with a confirmed IC-OR per investigator, was defined as the time from the date of first dose to the first documentation of objective intra-cranial response (CR or PR) which is subsequently confirmed. For participants whose IC-OR proceeds from PR to CR, the onset of PR was taken as the onset of response. CR: disappearance of all target and non-target lesions. PR: at least 30 % decrease in sum of diameters of target, taking as reference baseline sum diameters.
Time Frame: as for outcome 15
Population: PPINV included all enrolled participants who took at least 1 dose of Lorlatinib and had CNS metastases at study entry (i.e. with lesions having disease site = brain) according to investigator. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Lorlatinib
Number analyzed (Participants) | 13
Months | 2.8 [1.3 to 15.3]

17. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in participant or clinical study participant, temporally associated with use of study intervention, whether or not considered related to study intervention. A TEAE was defined as any event that occurs for first time during on-treatment period or AEs that were observed prior to start of study treatment but increased in severity during on-treatment period (defined as time from first dose of study treatment through end of safety follow-up period, ie at least 28 days, and no more than 35 days after discontinuation of treatment, or start of new anti-cancer therapies [follow up systemic therapy, follow up radiation therapy or follow-up surgery], whichever occurs first). Adverse events occurring on same day as first dose of study treatment were also considered to have occurred during the on-treatment period.
Time Frame: From first dose of the study treatment (Day 1) maximum up to 28-35 days after last dose of study drug or the new anti-cancer therapy date, whichever is earlier (maximum treatment exposure up to 43.78 months)
Population: Safety analysis set included all enrolled participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Participants | 69 [1.3 to 15.3]

18. Secondary Outcome: Number of Participants With Treatment-Related TEAEs
Description: An AE was any untoward medical occurrence in participant or clinical study participant, temporally associated with use of study intervention, whether or not considered related to study intervention. A TEAE was defined as any event that occurs for first time during on-treatment period or AEs that were observed prior to start of study treatment but increased in severity during on-treatment period (defined as time from first dose of study treatment through end of safety follow-up period, ie at least 28 days, and no more than 35 days after discontinuation of treatment, or start of new anti-cancer therapies [follow up systemic therapy, follow up radiation therapy or follow-up surgery], whichever occurs first). Adverse events occurring on same day as first dose of study treatment were also considered to have occurred during the on-treatment period. An AE was considered treatment related if investigator considered event related to study drugs or the information was unknown.
Time Frame: as for outcome 17
Population: Safety analysis set included all enrolled participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Participants | 64 [1.3 to 15.3]

19. Secondary Outcome: Number of Participants With Maximum Grade 3 or 4 TEAEs by National Cancer Institute Common Terminology Criteria for AEs [NCI CTCAE] v.4.03
Description: An AE was any untoward medical occurrence in participant or clinical study participant, temporally associated with use of study intervention, whether or not considered related to study intervention. A TEAE was defined as any event that occurs for first time during on-treatment period or AEs that were observed prior to start of study treatment but increased in severity during on-treatment period (defined as time from first dose of study treatment through end of safety follow-up period, ie at least 28 days, and no more than 35 days after discontinuation of treatment, or start of new anti-cancer therapies, whichever occurs first). Adverse events occurring on same day as first dose of study treatment were also considered to have occurred during the on-treatment period. TEAEs were graded according to NCI CTCAE v4.03 as grade 3= severe AE and grade 4= life threatening consequences; urgent intervention indicated.
Time Frame: as for outcome 17
Population: Safety analysis set included all enrolled participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Participants | 28 [1.3 to 15.3]

20. Secondary Outcome: Number of Participants With Maximum Grade 3 or 4 Treatment-Related AEs
Description: An AE was any untoward medical occurrence in participant or clinical study participant, temporally associated with use of study intervention, whether or not considered related to study intervention. An AE was considered treatment related if investigator considered event related to study drugs or the information was unknown. TEAEs were graded according to CTCAE v4.03 as grade 3= severe AE and grade 4= life threatening consequences.
Time Frame: as for outcome 17
Population: Safety analysis set included all enrolled participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Participants | 19 [1.3 to 15.3]

21. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs)
Description: A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions) or resulted in congenital anomaly/birth defect or was considered an important medical event. TESAEs were defined as any event that occurs for first time during on-treatment period or SAEs that were observed prior to start of study treatment but increased in severity during on-treatment period (defined as time from first dose of study treatment through end of safety follow-up period, ie at least 28 days, and no more than 35 days after discontinuation of treatment, or start of new anti-cancer therapies, whichever occurs first).
Time Frame: as for outcome 17
Population: Safety analysis set included all enrolled participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Participants | 23 [1.3 to 15.3]

22. Secondary Outcome: Number of Participants With Treatment-Related TESAEs
Description: SAE was any untoward medical occurrence at any dose that: resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions) or resulted in congenital anomaly/birth defect or was considered an important medical event. TESAEs were defined as any event that occurs for first time during on-treatment period or SAEs that were observed prior to start of study treatment but increased in severity during on-treatment period (defined as time from first dose of study treatment through end of safety follow-up period, ie at least 28 days, and no more than 35 days after discontinuation of treatment/ start of new anti-cancer therapies, whichever occurs first). SAE was considered treatment related if investigator considered event related to study drugs or information was unknown.
Time Frame: as for outcome 17
Population: Safety analysis set included all enrolled participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Lorlatinib
Number analyzed (Participants) | 71
Participants | 1 [1.3 to 15.3]

ADVERSE EVENTS:
Time Frame: From first dose of the study treatment (Day 1) maximum up to 28-35 days after last dose of study drug or the new anti-cancer therapy date, whichever is earlier (maximum treatment exposure up to 43.78 months)
Description: Safety analysis set. Same event may appear as both non-SAE and SAE. What is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. All-cause mortality: number of deaths are reported from Day 1 of the study up to 28-35 days post last dose and deaths which occurred after 28-35 days post last dose of study drug are also included.
Groups:
- Lorlatinib 100mg: Participants received Lorlatinib 100 mg (25 mg*4 tablets) orally QD in 21-day cycles. Participants continued to receive study treatment until objective disease progression, unacceptable toxicity, participant refusal, lost to follow up or death, whichever occurred first.
Arm/Group | Lorlatinib 100mg
All-Cause Mortality (participants affected / at risk) | 20/71
Serious Adverse Events (participants affected / at risk) | 23/71
Other Adverse Events (participants affected / at risk) | 66/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lorlatinib 100mg (N=71)
Right ventricular dysfunction (Cardiac disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
General physical health deterioration (General disorders) | 1
COVID-19 (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pneumonia viral (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Cranial nerve disorder (Nervous system disorders) | 1
Guillain-Barre syndrome (Nervous system disorders) | 1
Intracranial pressure increased (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lorlatinib 100mg (N=71)
Anaemia (Blood and lymphatic system disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 6
Asthenia (General disorders) | 14
Fatigue (General disorders) | 5
Oedema (General disorders) | 6
Oedema peripheral (General disorders) | 26
Pyrexia (General disorders) | 12
COVID-19 (Infections and infestations) | 8
Alanine aminotransferase increased (Investigations) | 4
Blood cholesterol increased (Investigations) | 19
Blood creatinine increased (Investigations) | 5
Blood glucose increased (Investigations) | 4
Blood triglycerides increased (Investigations) | 16
SARS-CoV-2 test positive (Investigations) | 5
Weight increased (Investigations) | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 24
Hyperlipidaemia (Metabolism and nutrition disorders) | 12
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 27
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/72/NCT04362072/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT04362072/SAP_001.pdf